CLINICAL TRIAL: NCT01720017
Title: The Impact of Airway Manikin Training on the Airtraq Avant and Wireless Monitor System Learning Curve in Airways With Predictors for Difficult Intubation
Brief Title: Impact of Manikin Training on Airtraq Avant Learning Curve in Predicted Difficult Airways
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty was encountered with the subjects completing their required 20 intubations in patients with at least one predictor of difficult intubation.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2012-0636
Record Dates: First submitted 2012-10-24; First posted 2012-11-01 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2014-05

CONDITIONS: Education; Training; Manikin
Keywords: Airtraq; laryngoscope; airway; difficult; training; manikin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inservice Training Only (Active Comparator): Inservice training will include review of a product information handout and a video demonstration. Specific attention will be given to (1) describing each system component and its operation, (2) attaching the wireless camera head and coordinating channel selection with the monitor, (3) turning on the Airtraq Avant light and device preparation for use, (4) Airtraq Avant insertion into the patient's mouth and advancement into the hypopharynx (deep in the throat) to obtain a view of the vocal cords, (5) use of standard lift and rotation movements to optimize the vocal cord view, (6) tracheal tube advancement through the vocal cords tracheal intubation, (7) standard methods for confirmation of correct tracheal tube placement, (8) tracheal tube removal from the Airtraq Avant and the Airtraq Avant removal from the patient's mouth, and (9) disposal of the disposable blade and cleaning of the reusable optics insert.
  Interventions: Other: Inservice Training
- Inservice and Manikin Training (Experimental): Study subjects in this group will receive the standard inservice training described above, as well as, preclinical manikin training on use of the Airtraq Avant and Wireless Monitor System in simulated difficult airway conditions (swollen tongue and cervical collar). During the preclinical manikin training, each subject will perform 10 intubations. Performance characteristics including attempts for successful Airtraq Avant insertion, glottic view obtained, ease of insertion, ease of tracheal intubation, time required for tracheal intubation, and attempts for successful tracheal intubation will be recorded for each intubation.
  Interventions: Other: Preclinical Manikin Training

INTERVENTIONS:
Other: Preclinical Manikin Training — During the preclinical manikin training, each subject will perform 10 intubations in a manikin with a difficult airway simulated by swelling the manikin tongue and placing it in a cervical collar.
  Arms: Inservice and Manikin Training
Other: Inservice Training — Inservice training will include review of a product information handout and a video demonstration.
  Arms: Inservice Training Only

SUMMARY:
The overall purpose of this study is to assess the impact of preclinical airway manikin training using the Airtraq Avant and Wireless Monitor System under simulated difficult airway conditions (c-collar and swollen tongue) on the clinical learning curve of using the device/system in airways with predictors for difficult intubation.

The investigators hypothesize that the clinical learning curve in airways with predictors for difficult intubation will be shorter for study subjects (operators) who undergo preclinical manikin training under simulated difficult airway conditions compared to Study subjects (operators) who do not receive this training. The clinical learning curve is characterized by procedure times and first attempt success rates on successive uses of the Airtraq Avant and Wireless Monitor System in patients with at least one predictor for difficult intubation.

DETAILED DESCRIPTION:
Tracheal intubation (placement of a breathing tube below the vocal cords into the trachea) is an essential skill for the anesthesia provider. Training on the use of new technology (i.e., procedural training), including video/optical laryngoscopy (e.g., the Airtraq Avant, Glidescope, and similar devices) usually occurs under the tutelage of learned practitioners, while caring for actual patients in the operating room, not during didactic sessions in a classroom. Although the use of airway trainers (manikins) has led to improved clinical learning curves for the use of some airway devices, it is not known if training on the use of the Airtraq Avant and Wireless Monitor System under simulated difficult airway conditions (c-collar and swollen tongue) will improve the learning curve of using the device/system clinically in in patients with at least one predictor of difficult intubation.

The specific aim of this study is to compare the clinical learning curve, characterized by procedure times and first attempt success rates on successive uses, of using the Airtraq Avant and Wireless Monitor System in patients with at least one predictor for diffcult intubation between anesthesia providers who receive preclinical airway manikin training under simulated difficult airway conditions (c-collar and swollen tongue) and those who do not. The subjects of this study are anesthesia providers enrolled in the study.

Secondary specific aims include assessing the impact of preclinical airway manikin training under simulated difficult airway conditions on glottic view grade, glottic view attainment maneuvers, ease of Airtraq Avant insertion, ease of tracheal tube insertion, mechanisms of tracheal tube insertion impediment, and perceived overall clinical usefulness in airways with predictors of difficult intubation.

ELIGIBILITY:
Inclusion Criteria:

* anesthesia providers (i.e., anesthesia residents, anesthetists, and staff anesthesiologists)

Exclusion Criteria:

* < 18 years of age
* non-english speaking
* unwilling to sign a study consent form
* related financially or otherwise to the Airtraq Avant manufacturer will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Intubation time | Within the first 3 minutes of 20 successive intubations.
  Repeated measure of intubation efficiency using the Airtraq Avant and Wireless Monitor System in airways with at least one predictor of difficult intubation, defined as the time from placing the videolaryngoscope into the patient's mouth to passage of the tracheal tube balloon below the vocal cords.

SECONDARY OUTCOMES:
First attempt success rate | Within the first 3 minutes of 20 successive intubations.
  Cumulative measure of intubation success on first attempt over 20 successive uses of the Airtraq Avant and Wireless Monitor System in airways with at least one predictor of difficult intubation, defined as the ability to place a tracheal tube below a patient's vocal cords on the first attempt without removing the videolaryngoscope from the patient's mouth.

OTHER OUTCOMES:
Glottic view grade | Within the first 3 minutes of 20 successive intubations
  Determined as the best view obtained when attempting to use the Airtraq Avant and Wireless Monitor System to pass a tracheal tube below a patient's vocal cords. Grade 1 = full view of vocal cords. Grade 2a = partial view of vocal cords. Grade 2b = no vocal cords seen. Arytenoids visible. Grade 3 = No view of the vocal cords or arytenoids. Anterior epiglottis visible. Grade 4 = Only soft tissue visible. No view of the periglottic structures, including the epiglottis, is present.
Ease of Airtraq Avant insertion Avant insertion | Within the first 3 minutes of 20 successive intubations
  Graded by the study subject on a 6-point Lickert scale (1 = easy, no difficulty; 6 = difficult, nearly impossible) when attempting to insert the Airtraq Avant into a patient's mouth.
Ease of tracheal intubation | Within the first 3 minutes of 20 successive intubations
  Graded by the study subject on a 6-point Lickert scale (1 = easy, no difficulty; 6 = difficult, nearly impossible) when attempting to pass a tracheal tube below a patient's vocal cords using the Airtraq Avant and Wireless Monitor System.
Mechanisms of tracheal tube insertion impediment | Within the first 3 minutes of 20 successive intubations
  Observational description of features causing impediments to tracheal tube insertion (e.g., tube hitting the epiglottis or tube hitting the arytenoid). Recorded by the study subject at the time of attempt at placing a tracheal tube below a patient's vocal cords using the Aitraq Avant and Wireless Monitor System.
Overall clinical usefulness | Within the first 3 minutes of 20 successive intubations
  Recorded as excellent, good, fair, or inadequate by the study subject when using the Airtraq Avant and Wireless Monitor System to place a tracheal tube below a patient's vocal cords.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Galgon, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States